CLINICAL TRIAL: NCT01140152
Title: Proteomic Analysis Reveals Innate Immune Activity In Intestinal Transplant Dysfunction
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: NIH T32 Human and Molecular Development Training Grant (Unknown)
Responsible Party: Anjuli Kumar, M.D./Principal Investigator, UCLA
Other Study IDs: 08-06-058-02A
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-02

CONDITIONS: Intestinal Transplant; Cellular Rejection
Keywords: intestinal transplantation; rejection; proteomics; innate immunity
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ostomy effluent
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No rejection: Intestinal transplant recipients with no evidence of biopsy proven rejection
- Rejection: Intestinal transplant recipients who had evidence of biopsy proven rejection

SUMMARY:
Many patients with intestinal failure require intestinal transplantation for survival. Currently, the gold standard for diagnosing acute cellular rejection (ACR) is histological examination of endoscopic biopsies, which are taken invasively and lack sensitivity. A non-invasive method of monitoring for ACR is needed.

DETAILED DESCRIPTION:
INTRODUCTION:

Intestinal transplantation (ITx) offers a potential means of survival for patients with intestinal failure who have developed life threatening complications. Approximately 200 ITx procedures are performed worldwide per year, with 2200 such procedures having been performed in total, two thirds of which have been in children. Overall, patient and graft survival rates have improved significantly over the past several years due to innovations in surgical techniques, immunosuppression and post-transplant management. One year patient survival rates approach 80-90% at experienced centers. Nonetheless, acute cellular rejection (ACR) continues to pose major challenges in these patients.

Currently, the gold standard for diagnosing ACR is histological examination of biopsy samples obtained at the time of endoscopy. Limitations include the fact that endoscopy is by definition invasive, costly, associated with risks of bleeding, infection, or perforation, and potentially inaccurate. ACR can present as a patchy process which may be missed by endoscopic surveillance up to 30% of the time. It also presents in a similar fashion to infection, leading to a diagnostic dilemma as to the optimal management of the patient. Such delays and inaccuracies in the diagnosis and management of ITx recipients have the potential to lead to patient and graft loss. New noninvasive techniques to monitor for ACR are clearly needed to continue to drive the field of ITx forward.

Proteomics allows the identification of proteins as possible biomarkers. Protein profiles can be easily detected in body fluids, making these protein combinations potentially innovative biomarkers useful in diagnosis or disease monitoring. Following protein and metabolite levels may prove to be an accurate screening tool for patients suspected of having ACR.

In this study, we use high-throughput proteomic analysis and candidate immunoassay protein detection of ostomy effluents to search in a non-invasive manner for molecular profiles of epithelial stress and innate immunity during ACR.

IMMUNOSUPPRESSION:

All patients are managed with tacrolimus-based triple immunosuppression. Our standard immunosuppression regimen includes induction with an interleukin-2 receptor antagonist such as daclizumab or basiliximab, versus rabbit antithymocyte globulin. Maintenance therapy consists of tacrolimus, corticosteroids, and mycophenolate mofetil. Target tacrolimus trough levels are 10-15 ng/mL. Sirolimus is used as a rescue agent and as part of a renal sparing regimen. ACR is diagnosed by histopathology and treated with high dose steroids. In patients with severe ACR, ATG is used as a rescue agent. In highly sensitized patients or patients suspected of antibody mediated rejection, a combination of plasmapheresis, Rituximab and IVIG is used.

INTESTINAL SURVEILLANCE:

Protocol biopsies of the transplanted intestine are obtained once weekly beginning postoperative day 7-14 for the first 3-4 weeks, then once every 2 weeks until 8 weeks after ITx. Endoscopy and biopsies are also obtained for clinical symptoms indicating abnormal allograft function. Multiple targeted biopsies are obtained, and paraffin-embedded sections stained with hematoxylin and eosin (H&E) are graded for ACR using standard rejection criteria by one of three UCLA gastrointestinal pathologists. Abnormal results prompt further endoscopic surveillance as indicated.

OSTOMY EFFLUENT COLLECTION AND PROTEOMIC EVALUATION:

Ostomy effluents are collected, immediately placed on ice, and batch processed at the UCLA High Throughput Clinical Proteomics mass spectrometry core laboratory. All samples are processed and analyzed in triplicate using MALDI mass spectrometry. MALDI-MS spectra are converted to text files, and preprocessed using an established protocol. The preprocessed MALDI data are then exported from SpecAlign and further analyzed in R.

ENZYME LINKED IMMUNOSORBENT ASSAY AND IMMUNOHISTOCHEMISTRY:

Human HNP 1-3 is quantified in duplicate processed protein samples by an ELISA kit following manufacturer's instructions (Cell Sciences, Canton, MA), using an HNP1-3 standard curve constructed for each plate. Protein concentrations are also determined for each test sample (BCA, Pierce Thermo Scientific, Rockford, IL), and HNP1-3 levels normalized to total protein (pg/mg).

For IHC, biopsy sections are deparaffinized, blocked for background peroxidase activity and goat antibody binding by standard methods, and stained with human anti-HNP 1-3 antibody (rabbit, 1:2000) or pre-immuned serum (rabbit, 1:2000) as negative control. The sections are further incubated with an anti-Rabbit IgG biotinylated secondary antibody and streptavidin-peroxidase conjugated tertiary antibody from the Vectastain Elite ABC kit (Vector Laboratories) according to the manufacturer's protocol, and developed by diaminobenzidine tetrahydrochloride (DAB) substrate solution (Pierce, Rockford, IL). For IHC quantitation, 10 crypts in three different fields on the biopsy slide are evaluated for evidence of significant defensin staining. The number of defensin positive crypts are counted and averaged.

LUMINEX:

An aliquot of processed ostomy effluent is used for Luminex evaluation, with the Bio-Rad human cytokine 17-plex assay according to the manufacturer's instructions (Bio-Rad, Hercules, CA). Data is acquired on a Bio-Plex 200 system and analyzed with associated software (Bio-Rad), and cytokine concentrations are normalized to protein concentration and log transformed.

ELIGIBILITY:
Inclusion Criteria:

* Intestinal transplant recipient
* Less than 8 weeks post transplant

Exclusion Criteria:

* Intestinal transplant recipients more than 8 weeks post transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Intestinal transplant recipients at UCLA, who are up to 8 weeks status-post transplant and are undergoing surveillance endoscopy or who present with elevated stool outputs with concern for acute rejection. Controls will consist of all primary ITx recipients of the same follow-up criteria who are undergoing surveillance biopsies but are at their baseline ostomy outputs.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evaluate levels of proteins and cytokines in ostomy effluent during episodes of rejection | first 8 weeks post transplant
  Protocol biopsies of the transplanted intestine are obtained during endoscopy and when clinical symptoms indicating abnormal allograft function are present. Biopsies were sent to pathology, where the pathologist determined if there was acute rejection.
  Ostomy effluent taken during times of endoscopy were subjected to MALDI and Luminex technology to look for any proteins or cytokines differentially expressed during rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Anjuli R Kumar, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States